CLINICAL TRIAL: NCT02931669
Title: What Does AAC Mean to You?: An Exploration of the Meaning and Value of AAC to Users and Stakeholders.(AAC: Augmentative and Alternative Communication)
Brief Title: Meaning, Value and Purpose of Augmentative and Alternative Communication (AAC)
Acronym: AAC
Status: Completed | Type: Observational
Sponsor: University of Dublin, Trinity College (Other)
Collaborators: National Health Service, United Kingdom (Other Government)
Responsible Party: Principal Investigator, Denise Abraham, Specialist Speech and Language Therapist (Severe and Complex Needs), University of Dublin, Trinity College
Other Study IDs: U Dublin TC; 200453 (Other: NHS - IRAS number)
Record Dates: First submitted 2016-10-11; First posted 2016-10-13 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Meaning, Value and Purpose of AAC

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Adult AAC users: Will be accessed via online forums to fill in online anonymous survey link
  Interventions: Other: Qualitative Descriptive Study
- Children who use AAC: Parents at local special schools will be given the opportunity for their child to participate in a face to face symbol based interview. They will give written consent and children's assent will also be obtained.
  Interventions: Other: Qualitative Descriptive Study
- Family members: The paper version of the survey will be distributed among parents at local special schools for them to fill in at home with their families. Online groups of families will also be sent the online survey link.
  Interventions: Other: Qualitative Descriptive Study
- Teachers: Teachers at local special schools will be given the paper survey forms. Online groups of teachers will receive the online link.
  Interventions: Other: Qualitative Descriptive Study
- Health Professionals: Online groups of health professionals will receive the online link
  Interventions: Other: Qualitative Descriptive Study

INTERVENTIONS:
Other: Qualitative Descriptive Study

SUMMARY:
The perception of disability has changed throughout history, and today, people who previously did not have a way to communicate are able to express themselves through Augmentative and Alternative Communication (AAC). However, the potential of AAC is not being fully realised and devices are often abandoned. It is therefore essential to hear the voice of those who use it and those who interact with them on a daily basis, in order to find out what the meaning, value and purpose of AAC is for them. This will support SLTs in directing intervention and establishing priorities, as well as in advocating for funding and acknowledging the voice of AAC users. The study uses a qualitative descriptive approach, using thematic analysis to establish emerging themes from surveys completed by AAC users, family members, health professionals, teachers, and face to face interviews with children who use AAC.

DETAILED DESCRIPTION:
Research indicates that AAC (Augmentative and Alternative Communication) has the potential to change the lives of many people with complex communication needs, but is often under-utilised and/or abandoned. Therefore, the research aims to investigate the meaning, value, and purpose of AAC for different stakeholder groups, as well as to what extent these are shared or unique? This information will support Speech and Language Therapists to understand the meaning, value, and purpose of AAC for key stakeholders, and therefore adapt intervention to meet these needs. It can also support families considering AAC in decision making. Participants can also benefit through reflecting on what AAC means to them. It is also an important part of evidence based practice to listen to the voice of the client and family.

A qualitative descriptive study is proposed, utilising thematic analysis. The study will be implemented using a survey which will be presented in different formats (paper/online/face-to-face) depending on the stakeholder. It will investigate the perceptions of people who use AAC, family members, teaching staff and health professionals who work with AAC users. Family members, adult AAC users, teachers and health professionals will receive a link to an online survey, distributed by professional groups and charities. Parents of children attending local special schools will be given paper copies of the survey. Face to face interviews with up to 5 children who use AAC will also be carried out at local special schools, following consent from the parents. Interviews will be conducted by a trained Speech and Language Therapist using symbols to support communication via a Talking Mats style approach,and children will be accompanied by an adult. It is estimated that interviews will last between 20 and 30 minutes.

Participants filling in the paper or online survey are encouraged to write as much or as little as they like; it is estimated that it will take around 10 minutes to complete, although others may spend longer.

ELIGIBILITY:
Inclusion Criteria:

* Those who use AAC (both children and adults), their family members and carers, and health professionals and teaching staff who work with AAC users.

Children who use AAC will be aged between 4 and 18 years of age. There is no age limit on other participants

Exclusion Criteria:

* Those who do not meet the inclusion criteria. No other exclusion criteria have been applied.

Max Age: 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: There are 5 potential groups as previously outlined: Adults who use AAC, children who use AAC, family members, teachers, and health professionals. Most will receive the online survey link through professional groups and online forums. The children who use AAC and some teachers and family members will be accessed through local special schools.
Sampling Method: Non-Probability Sample
Enrollment: 189 (Actual)
Dates: Start 2016-10; Primary Completion 2017-09-17 (Actual); Study Completion 2017-09-17 (Actual)

PRIMARY OUTCOMES:
Thematic Analysis of Survey Data | 08/2017

CONTACTS AND LOCATIONS:
Locations (1):
- Trinity College Dublin, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No